CLINICAL TRIAL: NCT00004154
Title: Randomized Chemoprevention Trial With 4-HPR (Fenretinide) in Superficial Bladder Cancer
Brief Title: Fenretinide in Treating Patients Who Have Undergone Surgery for Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000067387; MDA-ID-95236; NCI-G99-1621; NCI-T98-0051; ID95-236 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenretinide (Experimental): Fenretinide (4-HPR) 200 mg orally every day for 12 months taken 25 out of every 28 days.
  Interventions: Drug: Fenretinide
- Placebo (Placebo Comparator): Placebo orally every day for 12 months, taken 25 out of every 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenretinide — 200 mg/day (two 100 mg capsules) for 25 days of 28 day cycle.
  Other Names: 4-HPR
  Arms: Fenretinide
Other: Placebo — Two placebo capsules for 25 days of 28 day cycle.
  Arms: Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether fenretinide is more effective than a placebo in preventing the recurrence of bladder cancer after surgery to remove the tumor.

PURPOSE: This randomized phase III trial is studying fenretinide to see how well it works compared to a placebo in treating patients who are at risk for recurrent bladder cancer following surgery to remove the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy, mechanism of action, and toxicity of fenretinide in patients at risk of recurrent superficial bladder cancer after complete resection of initial tumor.
* Determine the treatment effects in modulating the expression of retinoid receptors, chromosomal abnormalities (numerical chromosomal abnormalities and DNA ploidy), apoptosis, and autocrine motility factor receptor (intermediate endpoint markers of recurrent disease) in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to lesion type (multifocal vs solitary). Patients are randomized to one of two treatment arms.

Patients receive either oral fenretinide or placebo on days 1-25. Courses repeat every 28 days for up to 1 year in the absence of disease progression, unacceptable toxicity, or development of a second primary cancer requiring therapy.

Patients are followed every 3 months for 15 months.

PROJECTED ACCRUAL: A total of 178 patients (89 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven solitary or multifocal superficial (stage Ta, grades 1-2) transitional cell carcinoma (TCC) of the bladder meeting 1 of the following criteria:

  * Newly diagnosed and no more than 4 weeks since resection
  * Secondary after being tumor free (including carcinoma in situ) for more than 12 months with no intravesical therapy within that 12 months OR
* Histologically proven Ta, T1, or Tis TCC of the bladder previously treated with Bacillus Calmette-Guerin (BCG).

  * Must have received 6 weeks of induction BCG followed by no evidence of disease by cystoscopy and cytology and then further treatment with 3 weekly doses of BCG.
* Visible tumor totally resected within 4 weeks prior to study entry and no further surgery, intravesical therapy, or systemic therapy planned
* No prostatic, prostatic urethral, or upper tract TCC involvement by the index tumor at resection
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod (Eastern Cooperative Oncology Group (ECOG)) 0-2

Life expectancy:

* At least 2 years

Hematopoietic:

* white blood count (WBC) greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 11.0 g/dL

Hepatic:

* serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) less than 1.5 times upper limit of normal (ULN)

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Triglyceride level less than 2.5 times ULN
* No other concurrent malignancy except nonmelanomatous skin cancer
* No other malignancy within the past 5 years unless currently disease free, at least 6 months since prior therapy, no current or planned active therapy, and expected disease-free survival at least 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after the study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent systemic biologic therapy

Chemotherapy:

* See Disease Characteristics
* No prior systemic cytotoxic chemotherapy for bladder cancer
* At least 1 year since prior cytotoxic chemotherapy for nonbladder cancer
* No concurrent systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the bladder
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 3 months since prior high-dose vitamin A (greater than 25,000 IU) or beta carotene (at least 30 mg/day)
* At least 3 months since prior retinoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 1998-07-30 (Actual); Primary Completion 2005-03-01 (Actual); Study Completion 2005-03-01 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of transitional cell carcinoma (TCC) | 1 year
  Recurrence rates is defined as proportion of participants who recur within one year of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anita L. Sabichi, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Sabichi AL, Lerner SP, Atkinson EN, Grossman HB, Caraway NP, Dinney CP, Penson DF, Matin S, Kamat A, Pisters LL, Lin DW, Katz RL, Brenner DE, Hemstreet GP 3rd, Wargo M, Bleyer A, Sanders WH, Clifford JL, Parnes HL, Lippman SM. Phase III prevention trial of fenretinide in patients with resected non-muscle-invasive bladder cancer. Clin Cancer Res. 2008 Jan 1;14(1):224-9. doi: 10.1158/1078-0432.CCR-07-0733. PMID 18172274